CLINICAL TRIAL: NCT02300194
Title: Topical Morphine for Analgesia in Pediatric Procedures. Clinical Trial Randomized, Double-blind, Placebo.
Brief Title: Randomized, Double-blind, Placebo, Controlled Cross Over Design Topical Morphine for Analgesia in Pediatric Procedures
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn by investigators
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HGNPE-157
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pain
Keywords: Pain management
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topic Morphine (Active Comparator): Use of topic morphine for treatment of procedure associated pain
  Interventions: Drug: Topic Morphine
- Placebo (Placebo Comparator): Use of topic hydrogel (placebo) for treatment of procedure associated pain
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topic Morphine — Topical application of a 0.1% morphine gel in patients undergo a procedure. It will be applied 30 minutes before the procedure and the first day every 4 hours. General basic sedation and systemic analgesia will give for all the patients. Efficacy of treatment will be measured with FLACC scale.
  Other Names: Morphine gel
  Arms: Topic Morphine
Drug: Placebo — Topical application of a placebo hydrogel in patients undergo a procedure. It will be applied 30 minutes before the procedure and the first day every 4 hours. General basic sedation and systemic analgesia will give for all the patients. Efficacy of treatment will be measured with FLACC scale.
  Other Names: Placebo hidrogel
  Arms: Placebo

SUMMARY:
Introduction:

Opioids, such as morphine, act at receptors in the central nervous system, but many studies have suggested direct action peripherally on opioid receptors in sensory neurons terminals, melanocytes, keratinocytes and fibroblasts. These receptors are stimulated when occurs inflammatory processes.

Hypothesis:

Treatment with topical morphine 0.1% applied 30 minutes before an invasive procedure, decreases pain in children.

Method:

A randomised double-blind parallel study to evaluate the effect of topical application of a 0.1% morphine gel in patients undergo a procedure. 22 patients in each group will be included. Randomly assigned to either the morphine gel or a placebo hydrogel, it will be applied 30 minutes before the procedure and the first day every 4 hours. General basic sedation and systemic analgesia will give for all the patients. Efficacy of treatment will be measured with "Face, Legs, Activity, Cry, Consolability scale" (FLACC scale).

DETAILED DESCRIPTION:
The use of an opioid such as morphine topical gel 30 minutes before a procedure would be effective in reducing pain in children. It has proven effective analgesic with minimal adverse effects, especially in children older than 6 months, and even its use is authorized in young children.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized children aged 1 month to 10 years, who needs a medical procedure over previously injured skin, associated with moderate-severe pain.

Exclusion Criteria:

* Refusal to participate

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | 4 hours
  Proportion of patients with a reduction in pain of least 2 point according to FLACC scale

CONTACTS AND LOCATIONS:
Overall Officials: María L Yazde-Puleio, MD, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de Niños Pedro de Elizalde, Buenos Aires, Argentina

REFERENCES:
- [Background] Garcia Roig C, Caprotta G, de Castro MF, Germ RM, Lagomarsino E. [Analgesia and sedation in pediatric procedures Part 1: general aspects, sedation scales and pain assessment]. Arch Argent Pediatr. 2008 Oct;106(5):429-34. doi: 10.1590/S0325-00752008000500010. No abstract available. Spanish. PMID 19030643
- [Background] Shavit I, Keidan I, Augarten A. The practice of pediatric procedural sedation and analgesia in the emergency department. Eur J Emerg Med. 2006 Oct;13(5):270-5. doi: 10.1097/00063110-200610000-00005. PMID 16969231
- [Background] Nielsen BN, Aagaard G, Henneberg SW, Schmiegelow K, Hansen SH, Romsing J. Topical morphine for oral mucositis in children: dose finding and absorption. J Pain Symptom Manage. 2012 Jul;44(1):117-23. doi: 10.1016/j.jpainsymman.2011.06.029. Epub 2012 Jun 1. PMID 22658469
- [Background] Heilmann S, Kuchler S, Schafer-Korting M. Morphine metabolism in human skin microsomes. Skin Pharmacol Physiol. 2012;25(6):319-22. doi: 10.1159/000342067. Epub 2012 Sep 8. PMID 22964846
- [Background] Ribeiro MD, Joel SP, Zeppetella G. The bioavailability of morphine applied topically to cutaneous ulcers. J Pain Symptom Manage. 2004 May;27(5):434-9. doi: 10.1016/j.jpainsymman.2003.09.011. PMID 15120772
- [Background] Watterson G, Howard R, Goldman A. Peripheral opioids in inflammatory pain. Arch Dis Child. 2004 Jul;89(7):679-81. doi: 10.1136/adc.2003.032003. PMID 15210505
- [Background] Nilsson S, Finnstrom B, Kokinsky E. The FLACC behavioral scale for procedural pain assessment in children aged 5-16 years. Paediatr Anaesth. 2008 Aug;18(8):767-74. doi: 10.1111/j.1460-9592.2008.02655.x. PMID 18613934
- See also: World Health Organization 2012 — https://apps.who.int/iris/handle/10665/77943